CLINICAL TRIAL: NCT05572866
Title: Before and After- Impact of COVID-19 Pandemic on Hepatobiliary and Pancreatic Surgical Services in Singapore: Retrospective Quantitative Study 2019-2022
Brief Title: Impact of COVID-19 Pandemic on Hepatopancreatobiliary Surgical Services in Singapore
Status: Completed | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ttshhpb
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: COVID-19; Surgery
MeSH Terms: conditions — COVID-19 | interventions — Pandemic Preparedness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 2019: No intervention will be carried out. The sum total of surgeries carried out during 2019 will be audited to see how the COVID-19 pandemic has impacted the surgical volume.
  Interventions: Other: COVID-19 pandemic
- 2020: No intervention will be carried out. The sum total of surgeries carried out during 2020 will be audited to see how the COVID-19 pandemic has impacted the surgical volume.
  Interventions: Other: COVID-19 pandemic
- 2021: No intervention will be carried out. The sum total of surgeries carried out during 2021 will be audited to see how the COVID-19 pandemic has impacted the surgical volume.
  Interventions: Other: COVID-19 pandemic
- 2022: No intervention will be carried out. The sum total of surgeries carried out during 2022 will be audited to see how the COVID-19 pandemic has impacted the surgical volume.
  Interventions: Other: COVID-19 pandemic

INTERVENTIONS:
Other: COVID-19 pandemic — To retrospectively review the surgical volume across 2019-2022 to see the impact of the COVID-19 pandemic.

SUMMARY:
This paper is intended to report our observational study in evaluating the impact of the COVID-19 pandemic on Tan Tock Seng Hospital hepatopancreatobiliary unit's surgical workload from January to June across 2019 to 2022, corresponding to the pre-pandemic baseline to its peak and the gradual normalization of hospital services as Singapore entered the transition phase to COVID-19 resilience.

DETAILED DESCRIPTION:
This paper is intended to report our observational study in evaluating the impact of the COVID-19 pandemic on Tan Tock Seng Hospital hepatopancreatobiliary unit's surgical workload from January to June across 2019 to 2022, corresponding to the pre-pandemic baseline to its peak and the gradual normalization of hospital services as Singapore entered the transition phase to COVID-19 resilience.

A comparative audit of the unit's surgical workload for the months of January-June across 2019 to 2022, which corresponded to pre-COVID-19, the height of the pandemic, and a gradual normalization of surgical services. Operations performed by the unit were collected from the surgeons' electronic case logs. These operations were sorted based on the Singapore Ministry of Health's table of surgical procedures, which assigns charge codes to different procedures. The retrospective data across the 4 years were compared and analysed.

No patient contact or identifiers were retrieved, stored or disseminated and thus exempt from ethics board review.

ELIGIBILITY:
Inclusion Criteria:

* all patients who underwent gallbladder, hernia, liver or pancreas resection surgeries during the periods of January to June of 2019/2020/2021/2022.

Exclusion Criteria:

* anyone who does not fall within the inclusion criteria

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent gallbladder, hernia, liver or pancreas resection surgeries during the periods of January to June of 2019/2020/2021/2022.
Sampling Method: Probability Sample
Enrollment: 1089 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of surgeries done under general anaesthesia by the hepatopancreatobiliary unit | 2019-2022
  Operations performed by the unit will be collected from the surgeons' electronic case logs. These operations will be sorted based on the Singapore Ministry of Health's table of surgical procedures, which assigns charge codes to different procedures. The retrospective data across the 4 years will be compared and analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Vishalkumar G Shelat, MMed, FRCS, Study Director — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.

REFERENCES:
- [Derived] Lim JSH, Lim ZY, Teo ZHT, Wang B, Tan YP, Junnarkar SP, Low JK, Huey CWT, Shelat V. Before and after COVID-19 pandemic: impact on hepatobiliary and pancreatic surgical services in a Singapore Tertiary Hospital. ANZ J Surg. 2023 Dec;93(12):2904-2909. doi: 10.1111/ans.18748. Epub 2023 Oct 27. PMID 37888881